CLINICAL TRIAL: NCT01099579
Title: A Prospective Single Arm, Open-label, International, Multicenter Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Atazanavir (ATV) Powder Boosted With Ritonavir (RTV) With an Optimized NRTI Background Therapy, in HIV Infected Pediatric Patients Greater Than or Equal to 3 Months to Less Than 6 Years. (Pediatric Atazanavir International Clinical Evaluation: the PRINCE I Study)
Brief Title: PRINCE: Study of Atazanavir (ATV)/Ritonavir (RTV)
Acronym: PRINCE1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI424-397; 2009-016361-28 (EudraCT Number)
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: HIV Infections
Keywords: HIV, Pediatric
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Atazanavir powder, 150 mg/Ritonavir oral solution, 80 mg (Experimental): Patients weighing 5 to <10 kg received atazanavir (ATV), 150-mg powder dosed in 50-mg packets, and ritonavir (RTV) oral solution, 80 mg. Stage 1: Initial dose was determined by patient's weight on the day of first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage. All of the mixture must have been consumed to obtain the full dose. The RTV oral solution was taken immediately before or after the ATV powder preparation. Stage 2: Patients who reached the age of 6 years or a weight of ≥25kg transitioned from the powder to the capsule formulation of ATV. Patients who weighed 15 to <20 kg received ATV, 150 mg with RTV, 100 mg; those who weighed 20 to <40 kg received ATV, 200 mg, and RTV, 100 mg; and those who weighed at least 40 kg received ATV, 300 mg with RTV, 100 mg. RTV capsules or tablets were ingested with food immediately before or after ATV intake.
  Interventions: Drug: Atazanavir powder; Drug: Ritonavir oral solution; Drug: Atazanavir capsules; Drug: Ritonavir capsules
- Atazanavir powder, 200 mg/Ritonavir oral solution, 80 mg (Experimental): Patients weighing 10 to <15 kg received ATV powder, 200 mg, dosed in 50-mg sachet packets and RTV oral solution, 80 mg. Stage 1: Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). All of the mixture must have been consumed to obtain the full dose. The RTV oral solution was taken immediately before or after the ATV powder preparation. Stage 2: Patients who reached the age of 6 years or a weight of ≥25kg transitioned from the powder to the capsule formulation of ATV. Patients who weighed 15 to <20 kg received ATV, 150 mg with RTV, 100 mg; those who weighed 20 to <40 kg received ATV, 200 mg, and RTV, 100 mg; and those who weighed at least 40 kg received ATV, 300 mg with RTV, 100 mg. RTV capsules or tablets were ingested with food immediately before or after ATV intake.
  Interventions: Drug: Atazanavir powder; Drug: Ritonavir oral solution; Drug: Atazanavir capsules; Drug: Ritonavir capsules
- Atazanavir powder, 250 mg/Ritonavir oral solution, 80 mg (Experimental): Patients weighing 15 to <25 kg received 250 mg of ATV powder dosed in 50-mg sachet packets, with 80 mg of RTV solution. Stage 1: Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). All of the mixture must have been consumed to obtain the full dose. The RTV oral solution was taken immediately before or after the ATV powder preparation. Stage 2: Patients who reached the age of 6 years or a weight of ≥25kg transitioned from powder to the capsule formulation of ATV. Patients who weighed 15 to <20 kg received ATV, 150 mg with RTV, 100 mg; those who weighed 20 to <40 kg received ATV, 200 mg, and RTV, 100 mg; and those who weighed at least 40 kg received ATV, 300 mg with RTV, 100 mg. RTV capsules or tablets were ingested with food immediately before or after ATV intake.
  Interventions: Drug: Atazanavir powder; Drug: Ritonavir oral solution; Drug: Atazanavir capsules; Drug: Ritonavir capsules

INTERVENTIONS:
Drug: Atazanavir powder — Powder, oral, dosed by weight. Participants who weighed 5 to <10 kg received atazanavir (ATV), 150 mg, and ritonavir (RTV), 80 mg; those who weighed 10 to <15 kg received ATV, 200 mg, and RTV, 80 mg; and those who weighed 15 to <25 kg received ATV, 250 mg, and RTV, 80 mg, once per day for 48 weeks or until pediatric indication is locally approved and participant meets requirements to receive appropriate formulation.
  Other Names: Reyataz; BMS-232632
Drug: Ritonavir oral solution — Oral solution, 80 mg/mL, once per day for 48 weeks or until pediatric indication is locally approved and participant meets requirements to receive appropriate formulation.
  Other Names: Norvir
Drug: Atazanavir capsules — Capsules, oral, dosed by weight in Stage 2. Patients who reached the age of 6 years or a weight of ≥25 kg transitioned from the powder to the capsule formulation of atazanavir (ATV). Patients who weighed 15 to <20 kg received ATV, 150 mg with RTV, 100 mg; those who weighed 20 to <40 kg received ATV, 200 mg, and RTV, 100 mg; and those who weighed at least 40 kg received ATV, 300 mg with RTV, 100 mg. RTV capsules or tablets were ingested with food immediately before or after ATV intake.
Drug: Ritonavir capsules — Oral, capsules, 100 mg, administered in Stage 2 with atazanavir capsules, dosed by weight.

SUMMARY:
The purpose of this study is to determine whether atazanavir powder combined with ritonavir is safe and well tolerated and produces appropriate drug exposure in children ≥3 months to <6 years of age.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed human immunodeficiency virus (HIV)-1 infection diagnosed by a positive virologic test result on 2 separate occasions by:

  * HIV DNA polymerase chain reaction
  * HIV RNA with values ≥1,000 copies/mL
  * Positive HIV enzyme-linked immunosorbent assay at ≥18 months of age, with confirmatory Western blot or indirect immunoflourescence antibody
* Infants and children of either sex, aged ≥3 months to <5 years and 6 months at time of first treatment, and weight >5 to <25 kg with any screening baseline plasma viral load
* Screening plasma viral load ≥1,000 copies/mL by Roche Amplicor® HIV RNA Assay
* Documented genotypic and phenotypic sensitivity at screening to ATV (fold change in susceptibility <2.2) and to at least 2 nucleoside reverse transcriptase inhibitors (NRTIs) approved in the infant's country
* Genotypic sensitivity at screening to atazanavir (ATV) and at least 2 NRTIs
* Antiretroviral (ARV) treatment-naive or ARV treatment-experienced. Treatment-experienced participants are defined by previous exposure to ARVs through either prior treatment for HIV infection or through postnatal treatment with ≥1 ARV for the prevention of mother to child transmission. For the purposes of this study, participants exposed to ARVs in utero or intrapartum may be included in the study but will be considered treatment naive. ATV-naive participants must have genotypic sensitivity at screening to ATV (fold change in susceptibility <2.2) and to both components of the local NRTI backbone. The NRTIs must have been approved for pediatric use at the local country level.

Key Exclusion Criteria:

* Experienced participants who received ATV or ATV/ritonavir (RTV) at any time prior to study enrollment or with a history of 2 or more protease inhibitor failures
* ARV-naïve or -experienced HIV-1 infected patients with contraindication to study medications syncope
* Family history of QTc interval syndrome, Brugada syndrome, right ventricular dysplasia, or a corrected QTc interval at screening of >440 ms
* One of the following cardiac rhythm abnormalities documented on screening electrocardiogram: 1st degree atrioventricular (AV) block as defined by protocol, type I 2nd degree AV block while awake, type II 2nd degree AV block at any time, complete AV block at any time, or age-adjusted heart rate <2nd percentile) History of pancreatitis, peripheral neuropathy, malignancy that requires systemic therapy, or any medical condition which, in the opinion of the investigator, added undue risk to trial participation
* Malabsorption syndrome
* Presence of a newly diagnosed HIV-related opportunistic infection or any medical condition requiring acute therapy at the time of enrollment
* Weight <5 or ≥25 kg at date of first dose (Day 1).
* >Grade 2 aspartate transaminase or alanine transaminase abnormalities
* Hypersensitivity to any component of the study medication formulations (ATV/RTV, or a locally prescribed NRTI with a pediatric indication)
* Infants and children of either gender <3 months or ≥5 years and 6 months at the time of first treatment.

Ages: 3 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2010-10-13 (Actual); Primary Completion 2012-10-04 (Actual); Study Completion 2017-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- Local Institution, São Paulo, São Paulo, Brazil
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Mexico (5):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Mérida, Yucatán
  - Local Institution, Oaxaca City
  - Local Institution, Puebla City
- Local Institution, Lima, Peru
- South Africa (5):
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Coronationville, Gauteng
  - Local Institution, Soweto, Gauteng
  - Local Institution, KwaKhangela, KwaZulu-Natal
  - Local Institution, Cape Town, Western Cape
- Local Institution, Bangkok, Thailand

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 82 pediatric patients were enrolled, and 56 received treatment. Reasons for not receiving treatment treated were: no longer met study criteria (23 patients), other reason (2 patients), and withdrew consent (1 patient).
Groups:
- Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg: Patients weighing 5 to <10 kg received atazanavir (ATV), 150-mg powder dosed in 50-mg sachet packets, and ritonavir (RTV) oral solution, 80 mg. Stage 1: Initial dose was determined by patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). If water was used, mixture must have been taken with food. The entire contents of the mixture must have been consumed to obtain the full dose. The ritonavir oral solution was taken immediately before or after the ATV powder preparation. Stage 2: Patients who reached the age of 6 years or a weight of 25 kg were transitioned to the capsule formulation of ATV. Those who weighed 15 to <20 kg received ATV, 150 mg, with RTV, 100 mg; those who weighed 20 to <40 mg received ATV, 200, with RTV, 100 mg; and those who weighed at least 40 mg received ATV, 300 mg, with RTV, 100 mg.
- Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg: Patients weighing 10 to <15 kg received ATV powder, 200 mg, dosed in 50-mg sachet packets and RTV oral solution, 80 mg. Stage 1: Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). If water was used, mixture must have been taken with food. All of the mixture must have been consumed to obtain the full dose. The RTV oral solution was taken immediately before or after the ATV powder preparation. Stage 2: Patients who reached the age of 6 years or a weight 25 kg were transitioned to the capsule formulation of ATV. Those who weighed 15 to <20 kg received ATV, 150 mg, with RTV, 100 mg; those who weighed 20 to <40 mg received ATV, 200, with RTV, 100 mg; and those who weighed at least 40 mg received ATV, 300 mg, with RTV, 100 mg.
- Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg: Patients weighing 15 to <25 kg received 250 mg of ATV powder dosed in 50-mg sachet packets, with 80 mg of RTV solution. Stage 1: Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). If water was used, mixture must have been taken with food. The entire contents of the mixture must have been consumed to obtain the full dose. The ritonavir oral solution was taken immediately before or after the ATV powder preparation. Stage 2: Patients who reached the age of 6 years or a weight 25 kg were transitioned to the capsule formulation of ATV. Those who weighed 15 to <20 kg received ATV, 150 mg, with RTV, 100 mg; those who weighed 20 to <40 mg received ATV, 200, with RTV, 100 mg; and those who weighed at least 40 mg received ATV, 300 mg, with RTV, 100 mg.
Period: Stage 1 (ATV Powder Formulation)
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Started | 21 | 19 | 16
Completed | 17 (Completed Stage 1) | 14 (Completed Stage 1) | 15 (Completed Stage 1)
Not Completed | 4 | 5 | 1
Not completed — Adverse Event | 4 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Poor compliance/noncompliance | 0 | 2 | 0
Period: Stage 2 (ATV Capsule)
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Started | 16 | 14 | 15
Completed | 10 | 9 | 9
Not Completed | 6 | 5 | 6
Not completed — No longer met study criteria | 2 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Poor/Non-Compliance | 2 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg: Patients weighing 5 to <10 kg received atazanavir (ATV), 150-mg powder dosed in 50-mg sachet packets, and ritonavir (RTV) oral solution, 80 mg. Stage 1: Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). If water was used, mixture must have been taken with food. The entire contents of the mixture must have been consumed to obtain the full dose. The ritonavir oral solution was taken immediately before or after the ATV powder preparation. Stage 2: Patients who reached the age of 6 years or a weight 25 kg were transitioned to the capsule formulation of ATV. RTV capsules or tablets were ingested with food immediately before or after ATV intake.
- Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg: Patients weighing 10 to <15 kg received ATV powder, 200 mg, dosed in 50-mg sachet packets and RTV oral solution, 80 mg. Stage 1: Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). If water was used, mixture must have been taken with food. All of the mixture must have been consumed to obtain the full dose. The RTV oral solution was taken immediately before or after the ATV powder preparation. Stage 2: Patients who reached the age of 6 years or a weight 25 kg were transitioned to the capsule formulation of ATV. Those who weighed 15 to 20 kg received ATV, 150 mg, with RTV, 100 mg, and those who weighed 20 to 40 mg received ATV, 200 mg with RTV,100 mg. RTV capsules or tablets were ingested with food immediately before or after ATV intake.
- Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg: Patients weighing 15 to <25 kg received 250 mg of ATV powder dosed in 50-mg sachet packets, with 80 mg of RTV solution. Stage 1: Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). If water was used, mixture must have been taken with food. The entire contents of the mixture must have been consumed to obtain the full dose. The ritonavir oral solution was taken immediately before or after the ATV powder preparation. Stage 2: Patients who reached the age of 6 years or a weight of 25 kg were transitioned to the capsule formulation of ATV. Those who weighed 20 to 40 mg received ATV, 200 mg, with RTV, 100 mg, and those who weighed at least 40 kg received ATV, 300 mg, with RTV, 100 mg. RTV capsules or tablets were ingested with food immediately before or after ATV intake.
- Total: Total of all reporting groups
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg | Total
Number analyzed (Participants) | 21 | 19 | 16 | 56
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.3 (4.05) | 35.4 (11.63) | 52.1 (10.49) | 29.6 (20.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 6 | 28
  Male | 11 | 7 | 10 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 0 | 0 | 1 | 1
  Not reported | 21 | 19 | 15 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 3 | 6 | 11
  Black/African American | 13 | 12 | 7 | 32
  Asian | 0 | 1 | 0 | 1
  Other | 6 | 3 | 3 | 12
Country [Count of Participants; unit: Participants]
  Chile | 1 | 2 | 3 | 6
  Mexico | 2 | 3 | 4 | 9
  Peru | 1 | 0 | 1 | 2
  South Africa | 17 | 13 | 8 | 38
  Thailand | 0 | 1 | 0 | 1
HIV RNA [Mean (Standard Deviation); unit: Log10 c/mL] | 4.77 (0.602) | 4.83 (0.268) | 4.18 (0.727) | 4.62 (0.617)
HIV RNA [Number; unit: c/mL]
  <30,000 c/mL | 3 | 2 | 9 | 14
  30,000 to 100,000 c/mL | 0 | 7 | 3 | 10
  >100,000 c/mL | 18 | 10 | 4 | 32
CD4 Count [Mean (Standard Deviation); unit: Cells/mm^3] | 1594.1 (897.19) | 1107.4 (643.25) | 661.1 (302.60) | 1192.6 (784.08)
CD4 Percent [Mean (Standard Deviation); unit: Percentage] | 25.4 (12.11) | 22.0 (9.35) | 27.5 (9.85) | 24.8 (10.61)
CD4 Percent [Count of Participants; unit: Participants]
  <15 | 2 | 2 | 1 | 5
  15 to <25 | 7 | 6 | 4 | 17
  >=25 | 7 | 6 | 6 | 19
  Not reported | 5 | 5 | 5 | 15
Prior Antiretroviral (ARV) Treatment Use [Count of Participants; unit: Participants] — ATV naive is defined as without prior exposure to ARV treatment; ARV experienced is defined as previous exposure to ARV drugs through prior treatment for HIV infection or through postnatal treatment with ≥1 ARVs for the prevention of mother-to-child-transmission in accordance with multiple international guidelines. Patients exposed to ARVs in utero or intrapartum were permitted in the study but were considered treatment naive.
  Participants
    ARV naive | 7 | 10 | 5 | 22
    ARV experienced | 14 | 9 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: From Day 1 to Week 48
Population: All participants who received at least 1 dose of active atazanavir powder.
Measure: Number; unit: Participants
Groups:
- Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg: Patients weighing 5 to <10 kg received atazanavir (ATV), 150-mg powder dosed in 50-mg sachet packets, and ritonavir (RTV) oral solution, 80 mg. Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). If water was used, mixture must have been taken with food. The entire contents of the mixture must have been consumed to obtain the full dose. The ritonavir oral solution was taken immediately before or after the ATV powder preparation.
- Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg: Patients weighing 10 to <15 kg received ATV powder, 200 mg, dosed in 50-mg sachet packets and RTV oral solution, 80 mg. Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). If water was used, mixture must have been taken with food. All of the mixture must have been consumed to obtain the full dose. The RTV oral solution was taken immediately before or after the ATV powder preparation.
- Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg: Patients weighing 15 to <25 kg received 250 mg of ATV powder dosed in 50-mg sachet packets, with 80 mg of RTV solution. Initial dose was determined by the patient's weight on the day of the first on-treatment study visit (Day 1). ATV dispersible powder was mixed with a small amount of food or beverage (water, milk, chocolate milk, liquid infant formula, applesauce, or yogurt). If water was used, mixture must have been taken with food. The entire contents of the mixture must have been consumed to obtain the full dose. The ritonavir oral solution was taken immediately before or after the ATV powder preparation.
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 21 | 19 | 16
Participants
  Deaths | 0 | 0 | 0
  SAEs | 5 | 2 | 4
  AEs leading to discontinuation | 4 | 1 | 0

2. Secondary Outcome: Percentage of Participants With HIV RNA Levels <50 c/mL and <400 c/mL at Week 48 by Treatment/Weight
Description: The definition of virologic success included HIV RNA levels <50 c/mL or 400 c/mL at the Week 48 analysis window. .
Time Frame: At Week 48
Population: Participants who received at least 1 dose of atazanavir and who did not switch to the capsule formulation at or before Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 21 | 19 | 14
Percentage of participants
  HIV RNA levels <50 c/mL | 47.6 | 68.4 | 71.4
  HIV RNA levels <400 c/mL | 66.7 | 73.7 | 85.7

3. Secondary Outcome: Percentage of Participants With HIV RNA Levels <50 c/mL and <400 c/mL at Week 48 by Prior Antiretroviral (ARV) Treatment Status
Description: The definition of virologic success included HIV RNA levels <50 c/mL or <400 c/mL at the Week 48 analysis.
Time Frame: From Day 1 to Week 48
Population: Participants who received at least 1 dose of atazanavir (ATV) and who did not switch to the ATV capsule formulation on or before Week 48
Measure: Number; unit: Percentage of participants
Groups:
- ARV-experienced: ARV-experienced participants had previous exposure to ARV drugs through prior treatment for HIV infection or through postnatal treatment with ≥1 ARVs for the prevention of mother-to-child-transmission in accordance with multiple international guidelines.
- ARV-naive: ARV-naive participants had no prior exposure to ARV treatment. Patients exposed to ARVs in utero or intrapartum were also considered treatment naive.
Arm/Group | ARV-experienced | ARV-naive
Number analyzed (Participants) | 20 | 34
Percentage of participants
  HIV RNA levels <50 c/mL | 56.3 | 68.2
  HIV RNA levels <400 c/mL | 65.6 | 86.4

4. Secondary Outcome: Mean Change From Baseline in HIV RNA Levels at Week 48 by Treatment/Weight
Description: Participants who received at least 1 dose of atazanavir (ATV) and had an HIV RNA measurement on ATV powder at did not switch to the capsule formulation before Week 48
Time Frame: From Baseline to Week 48
Population: Participants who received at least 1 dose of atazanavir and who had HIV RNA while taking atazanavir powder at Week 48
Measure: Mean (Standard Error); unit: Log10 c/mL
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 17 | 15 | 13
Log10 c/mL | -2.61 (0.3111) | -2.93 (0.1678) | -2.40 (0.2412)

5. Secondary Outcome: Mean Change From Baseline in HIV RNA Levels at Week 48 by Prior Antiretroviral (ARV) Treatment Status
Time Frame: From Baseline to Week 48
Population: Participants who received at least 1 dose of atazanavir (ATV) and who had an HIV RNA measurement on ATV powder at Week 48
Measure: Mean (Standard Error); unit: Log10 c/mL
Arm/Group | ARV-experienced | ARV-naive
Number analyzed (Participants) | 34 | 22
Log10 c/mL | -2.53 (0.2452) | -2.81 (0.1296)

6. Secondary Outcome: CD4 Cell Count Changes From Baseline at Week 48 by Treatment/Weight
Time Frame: From Baseline to Week 48
Population: Participants who received at least 1 dose of atazanavir (ATV) and who had CD4 at baseline and Week 48 while taking ATV powder
Measure: Mean (Standard Error); unit: Cells/mm^3
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 13 | 11 | 5
Cells/mm^3 | 550.1 (285.24) | 225.3 (198.34) | 373.8 (68.83)

7. Primary Outcome: Number of Participants With Laboratory Test Results With Worst Toxicity of Grade 3-4
Description: ALT=alanine aminotransferase; SGPT=serum glutamic-pyruvic transaminase; AST=aspartate aminotransferase; SGOT=serum glutamic-oxaloacetic transaminase; ULN=upper limit of normal. Grading by the National Institute of Health Division of AIDs and World Health Organization criteria. Hemoglobin (g/dL): Grade (Gr)1=9.5-11.0; Gr 2=8.0-9.4; Gr 3=6.5-7.9; Gr 4=<6.5. Neutrophils, absolute (/mm^3): Gr 1=>=1000-<1500; Gr 2= >=750-<1000; Gr 3=>=500-<750; Gr 4=<500. ALT/SGPT (*ULN): Gr 1=1.25-2.5; Gr 2=2.6-5; Gr 3=5.1-10; Gr 4=>10. AST/SGOT (*ULN): Gr 1=1.25-2.5; Gr 2=2.6-5; Gr 3=5.1-10; Gr 4=>10. Alkaline phosphatase(*ULN): Gr 1=1.25-2.5; Gr 2=2.6-5: Gr 3=5.1-10; Gr 4=>10. Total bilirubin (*ULN): Gr 1=1.1-1; Gr 2=1.6-2.5; Gr 3=2.6-5; Gr 4=>5. Amylase (*ULN): Gr 1=1.10-39; Gr 2=1.40-2; Gr 3=2.10-5.0; Gr 4=>5.0. Lipase (*ULN): Gr 1=1.10-1.39: Gr 2=1.40-2; Gr 3=2.10-5.0; Gr 4=>5.0. Uric acid (mg/dL): Gr 1=7.5-10.0; Gr 2=10.1-12.0; Gr 3=12.1-15.0; Gr 4=>15.
Time Frame: After Day 1 to Week 48
Population: All participants who received at least 1 dose of atazanavir; n=number of evaluable participants.
Measure: Number; unit: Participants
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 21 | 19 | 16
Participants
  Hemoglobin (n=20, 17, 15) | 2 | 3 | 0
  Neutrophils, absolute (n=20, 17, 15) | 3 | 2 | 0
  ALT/SGPT (n=20, 18, 15) | 5 | 0 | 1
  AST/SGOT (n=20, 18, 15) | 1 | 0 | 0
  Alkaline phosphatase (n=20, 18, 15) | 0 | 1 | 0
  Total bilirubin (n=20, 18, 15) | 2 | 0 | 3
  Amylase (n=20, 18, 15) | 8 | 5 | 1
  Lipase (n=20, 18, 15) | 0 | 1 | 1
  Uric acid n=20, 18, 15) | 0 | 0 | 1

8. Primary Outcome: Electrocardiogram Changes From Baseline in PR Interval, QTC Bazett, and QTC Fridericia at Week 48
Description: Electrocardiogram parameters were measured at baseline for QTC Bazett, QTC Fridericia, and PR interval. The mean change from baseline at week 48 is reported by arm in milliseconds.
Time Frame: From Baseline to Week 48
Population: All participants who received at least 1 dose of atazanavir and were evaluable
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 17 | 15 | 13
Milliseconds
  PR Interval | 4.9 (21.80) | 12.0 (8.04) | 6.2 (8.54)
  QTC Bazett | 1.7 (17.73) | -3.2 (21.78) | -4.2 (13.02)
  QTC Fridericia | 7.9 (18.36) | 13.2 (18.92) | 4.8 (11.49)

9. Primary Outcome: Number of Participants With Centers for Disease Control (CDC) Class C AIDS Events
Description: CDC Class C events are AIDS-defining events that include recurrent bacterial pneumonia (>=2 episodes in 12 months); candidiasis of the bronchi, trachea, lungs, or esophagus; invasive cervical carcinoma; disseminated or extrapulmonary coccidioidomycosis; extrapulmonary cryptococcosis; chronic intestinal cryptosporidiosis (>1 month); cytomegalovirus disease; HIV-related encephalopathy; herpes simplex: chronic ulcers, or bronchitis, pneumonitis, or esophagitis; disseminated or extrapulmonary histoplasmosis; chronic intestinal isosporiasis; Kaposi sarcoma; immunoblastic or primary brain Burkitt lymphoma; mycobacterium avium complex, kansasii, or tuberculosis; mycobacterium, other species; Pneumocystis carinii pneumonia; progressive multifocal leukoencephalopathy; Salmonella septicemia; recurrent toxoplasmosis of brain; HIV wasting syndrome (involuntary weight loss >10% of baseline body weight) with chronic diarrhea or chronic weakness and documented fever for ≥1 month.
Time Frame: From Day 1 to Week 48
Measure: Number; unit: Participants
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 21 | 19 | 16
Participants | 1 | 1 | 0

10. Secondary Outcome: CD4 Cell Count Changes From Baseline at Week 48 by Prior Antiretroviral (ARV) Treatment Status
Time Frame: From Baseline to Week 48
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Cells/mm^3
Arm/Group | ARV-experienced | ARV-naive
Number analyzed (Participants) | 34 | 22
Cells/mm^3 | 437.9 (253.123) | 352.1 (152.600)

11. Secondary Outcome: Mean CD4 Percent Changes From Baseline at Week 48 by Treatment/Weight
Time Frame: From Baseline to Week 48
Population: Participants who received at least 1 dose of atazanavir (ATV) and who had CD4 percent at baseline and Week 48 while taking ATV powder
Measure: Mean (Standard Error); unit: Percentage of lymphocytes
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 14 | 12 | 6
Percentage of lymphocytes | 6.1 (1.56) | 7.3 (2.26) | 8.8 (1.14)

12. Secondary Outcome: Mean CD4 Percent Changes From Baseline at Week 48 by Antiretroviral (ARV) Treatment Status
Time Frame: From Baseline to Week 48
Population: as for outcome 11
Measure: Mean (Standard Error); unit: Percentage of lymphocytes
Arm/Group | ARV-experienced | ARV-naive
Number analyzed (Participants) | 34 | 22
Percentage of lymphocytes | 4.3 (1.316) | 9.8 (1.496)

13. Secondary Outcome: Number of Participants Who Acquired Phenotypic Resistance to Atazanavir or Atazanovir/Ritonavir
Description: Criteria for resistance testing= meeting at least 1 of the following: <1 log10 drop from baseline in HIV RNA level by Week 16 and confirmed by a second HIV RNA level; an HIV RNA level >200 copies/mL after Week 24, confirmed by a second HIV RNA level; repeated HIV RNA levels ≥50 copies/mL after Week 48; an HIV RNA level ≥400 copies/mL confirmed by a second HIV RNA level of ≥400 copies/mL at any time in a participant who had previously achieved a plasma HIV RNA level <50 copies/mL; or discontinued due to lack of efficacy. Virologic failure was defined as an incomplete virologic response to therapy or as a viral rebound after the achievement of virologic suppression. The phenotypic resistance to a drug is defined as a fold change (ie, ratio of the 50% inhibitory concentration [IC50] of the clinical isolate to the IC50 of the reference strain) greater than the cut-off for reduced susceptibility.
Time Frame: After Day 1 to Week 48
Population: Participants who met the criteria for virologic failure
Measure: Number; unit: Participants
Arm/Group | ARV-experienced | ARV-naive
Number analyzed (Participants) | 6 | 8
Participants
  Atazanavir | 0 | 0
  Ritonavir | 0 | 0

14. Secondary Outcome: Maximum Observed Concentration (Cmax) and Minimum Observed Concentration (Cmin) of Atazanavir and Ritonavir
Time Frame: At Week 2 at Hour 0 predose and at Hours 1.5, 2.5, 4, 6, 8, 12, and 24 postdose
Population: All participants who had received study drug and had adequate pharmacokinetic profiles (n=number evaluable)
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 20 | 18 | 15
ng/mL
  Atazanavir Cmax | 4131 [1110 to 9660] | 5197 [390 to 15000] | 6172 [3560 to 10400]
  Atazanavir Cmin | 336 [11.4 to 1330] | 572 [11.2 to 4870] | 698 [238 to 2410]
  Ritonavir Cmax (n=19, 18, 15) | 2919 [188 to 9160] | 2634 [163 to 17700] | 1838 [582 to 4960]
  Ritonavir Cmin (n=18, 16, 15) | 41.8 [12.7 to 311] | 143 [14.2 to 1610] | 51.0 [9.0 to 468]

15. Secondary Outcome: Area Under the Concentration Curve (in 1 Dosing Interval From Time 0 to 24 Hours Post Observed Dose) (AUC[TAU])of Atazanavir and Ritonavir
Time Frame: At Week 2 at Hour 0 predose and at Hours 1.5, 2.5, 4, 6, 8, 12, and 24 postdose
Population: All participants who had received study drug and had adequate pharmacokinetic profiles (n=number evaluable)
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 20 | 18 | 15
ng*h/mL
  AUC(TAU) Atazanavir | 32503 [10441 to 94352] | 50305 [6697 to 189971] | 61485 [31599 to 117171]
  AUC(TAU) Ritonavir (n=19, 18, 15) | 17439 [1322 to 56864] | 20510 [971 to 229777] | 13640 [3376 to 40806]

16. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Atazanavir and Ritonavir
Time Frame: At Week 2 at Hour 0 predose and at Hours 1.5, 2.5, 4, 6, 8, 12, and 24 postdose
Population: All participants who had received study drug and had adequate pharmacokinetic profiles (n=number evaluable)
Measure: Median (Full Range); unit: Hours
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 20 | 18 | 15
Hours
  Tmax Atazanavir | 1.58 [1.40 to 12.0] | 1.97 [1.00 to 6.00] | 4.0 [1.5 to 6.0]
  Tmax Ritonavir | 1.8 [1.3 to 11.9] | 2.9 [1.0 to 8.0] | 4.0 [1.5 to 6.0]

17. Secondary Outcome: Apparent Total Body Clearance (CLT/F) of Atazanavir and Ritonavir
Description: Calculated as dose divided by AUC(TAU). AUC(TAU)=area under the concentration-time curve in 1 dosing interval from time 0 to 24 hours post observed dose.
Time Frame: At Week 2
Population: All participants who had received study drug and had adequate pharmacokinetic profiles (n=number evaluable)
Measure: Geometric Mean (Full Range); unit: L/h
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 20 | 18 | 15
L/h
  CLT/F Atazanavir | 4.61 [1.6 to 14.4] | 3.98 [1.1 to 29.9] | 4.07 [2.1 to 7.9]
  CLT/F Ritonavir (n=19, 18, 15 | 4.59 [1.4 to 60.5] | 3.90 [0.3 to 82.4] | 5.87 [2.0 to 23.7]

18. Secondary Outcome: Apparent Total Body Clearance Per Body Weight (CLT/F) Per Kilogram of Atazanavir and Ritonavir
Description: Calculated as CLT/F divided by body weight
Time Frame: At Week 2
Population: All participants who had received study drug and had adequate pharmacokinetic profiles (n=number evaluable)
Measure: Geometric Mean (Full Range); unit: L/h per kilogram
Arm/Group | Atazanavir Powder, 150 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 200 mg/Ritonavir Oral Solution, 80 mg | Atazanavir Powder, 250 mg/Ritonavir Oral Solution, 80 mg
Number analyzed (Participants) | 20 | 18 | 15
L/h per kilogram
  CLT/F per kilogram Atazanavir | 0.65 [0.2 to 1.8] | 0.32 [0.1 to 2.6] | 0.24 [0.1 to 0.5]
  CLT/F per kilogram Ritonavir (n=19, 18, 15) | 0.65 [0.2 to 7.5] | 0.32 [0.04 to 5.9] | 0.35 [0.1 to 1.4]

ADVERSE EVENTS:
Time Frame: From Day 1 to Week 48
Arm/Group | B/L Weight 5 to Less Than 10 kg | B/L Weight 10 to Less Than 15 kg | B/L Weight 15 to Less Than 25 kg
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19 | 0/16
Serious Adverse Events (participants affected / at risk) | 7/21 | 5/19 | 5/16
Other Adverse Events (participants affected / at risk) | 21/21 | 18/19 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/L Weight 5 to Less Than 10 kg (N=21) | B/L Weight 10 to Less Than 15 kg (N=19) | B/L Weight 15 to Less Than 25 kg (N=16)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Lymphadenitis bacterial (Infections and infestations) | 1 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Electrocardiogram qt prolonged (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/L Weight 5 to Less Than 10 kg (N=21) | B/L Weight 10 to Less Than 15 kg (N=19) | B/L Weight 15 to Less Than 25 kg (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Basophilia (Blood and lymphatic system disorders) | 1 | 1 | 1
Basophilopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 4 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Monocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 3
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 2
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 4 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 6 | 7
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1 | 0
Tongue geographic (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 9 | 8 | 4
Asthenia (General disorders) | 0 | 0 | 2
Local swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 7 | 5
Hepatomegaly (Hepatobiliary disorders) | 4 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 4
Jaundice (Hepatobiliary disorders) | 1 | 3 | 2
Ocular icterus (Hepatobiliary disorders) | 2 | 1 | 1
Acarodermatitis (Infections and infestations) | 6 | 0 | 1
Bacteriuria (Infections and infestations) | 1 | 1 | 1
Bronchitis (Infections and infestations) | 2 | 4 | 2
Candida nappy rash (Infections and infestations) | 5 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 2 | 1
Ear infection (Infections and infestations) | 1 | 1 | 0
Enterobiasis (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 2 | 1 | 0
Gastroenteritis (Infections and infestations) | 9 | 5 | 2
Helminthic infection (Infections and infestations) | 5 | 2 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 4 | 2 | 2
Influenza (Infections and infestations) | 3 | 1 | 2
Lice infestation (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 3 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1 | 5
Oral candidiasis (Infections and infestations) | 9 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 2
Otitis externa (Infections and infestations) | 3 | 3 | 1
Otitis media (Infections and infestations) | 8 | 4 | 4
Otitis media acute (Infections and infestations) | 3 | 2 | 2
Otitis media chronic (Infections and infestations) | 3 | 1 | 2
Parasitic gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 5 | 4 | 4
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 2
Pneumonia (Infections and infestations) | 4 | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Rhinitis (Infections and infestations) | 1 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 1
Tinea capitis (Infections and infestations) | 4 | 2 | 2
Tinea faciei (Infections and infestations) | 0 | 0 | 1
Tinea infection (Infections and infestations) | 1 | 1 | 3
Tonsillitis (Infections and infestations) | 7 | 2 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 6 | 5
Urinary tract infection (Infections and infestations) | 6 | 2 | 0
Varicella (Infections and infestations) | 2 | 1 | 1
Viral rash (Infections and infestations) | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 4 | 8 | 4
Vulvovaginal candidiasis (Infections and infestations) | 1 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 5 | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scar (Injury, poisoning and procedural complications) | 1 | 2 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Amylase increased (Investigations) | 2 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood sodium increased (Investigations) | 0 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 1
Crystal urine present (Investigations) | 0 | 1 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 2 | 1 | 0
Urinary sediment present (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 4 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 3 | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 3
Enuresis (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 6 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 7 | 4 | 1
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pityriasis alba (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Physical assault (Social circumstances) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.